CLINICAL TRIAL: NCT07309380
Title: Double-blinded Placebo-controlled Multi-center Phase III Clinical Trial of Hepalatide in Patients With Chronic Hepatitis D
Brief Title: Phase III Clinical Trial of Hepalatide in Patients With Chronic Hepatitis D
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai HEP Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: L47-HD-II/III-01
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Hepatitis D, Chronic
Keywords: hepalatide; L47
MeSH Terms: conditions — Hepatitis D, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Placebo Comparator): placebo of L47, sc,qd
  Interventions: Drug: Placebo of Hepalatide
- Group B (Experimental): hepalatide 2.1mg, sc, qd, Continuous treatment for 48 weeks
  Interventions: Drug: Hepalatide 2.1mg

INTERVENTIONS:
Drug: Hepalatide 2.1mg — Continuous treatment with hepalatide 2.1mg sc, qd, for 48 weeks
  Other Names: L47; HLT
  Arms: Group B
Drug: Placebo of Hepalatide — Continuous treatment with placebo of hepalatide for 48 weeks
  Arms: Group A

SUMMARY:
This study adopts a multicenter, randomized, double-blind, placebo-parallel controlled design to evaluate the efficacy and safety of L47 in the treatment of chronic hepatitis D.

A total of 150 subjects are planned to be enrolled. After passing the screening, they will be randomly assigned to the L47 group or the placebo group at a ratio of 2:1, with liver cirrhosis and subjects' regional distribution as stratification factors. The two groups will receive hepratide (2.1 mg/day) or placebo, respectively. Upon completion of the 48-week double-blind treatment phase, all subjects in each group can enter the open-label treatment follow-up phase, where they may voluntarily choose to receive L47 (2.1 mg/day) treatment or undergo follow-up observation only, until week 144.

Subjects who discontinue treatment prematurely during the trial may also enter the open-label treatment follow-up phase.

An interim analysis will be conducted after the subjects complete 24 weeks of trial treatment, with the comprehensive response rate at week 24 as the primary endpoint. The analysis will be performed by an independent statistical team. And the interim analysis results will be reviewed by the Independent Data Monitoring Committee (IDMC) .

All subjects will complete the 48-week double-blind clinical trial. Throughout the entire study period, the safety of subjects will be closely monitored and evaluated, including the monitoring of adverse events (AEs) and other safety indicators.

ELIGIBILITY:
Inclusion Criteria:

* Positive HBsAg or HBV DNA for at least 6 months (diagnosed as chronic hepatitis B), with stable nucleos(t)ide analogue (NA) treatment for ≥3 months prior to screening and documented HBV DNA suppression;
* Positive anti-HDV antibody (IgG and/or IgM) and at least two quantifiable HDV RNA measurements ≥3 months apart, with quantifiable HDV RNA at enrollment;
* 1×ULN< ALT<10×ULN；
* No plan for pregnancy within 2 years; female subjects must not be pregnant or lactating, and all subjects must agree to use effective contraception during treatment and for 3 months after the last dose;
* No participation in other clinical trials within 3 months prior to screening;
* Good compliance with the study protocol;
* Ability to understand and willingness to sign the informed consent form (ICF).

Exclusion Criteria:

* Child-Pugh class C or Child-Pugh score ≥10;
* Subjects with any of the following conditions:

  1. History of severe decompensated liver disease, including moderate to severe ascites (grade 2 or 3), hepatic encephalopathy, gastrointestinal variceal bleeding, hepatorenal syndrome, etc., with an expected survival of less than 2 years;
  2. History of severe cardiac disease (including unstable or uncontrolled heart disease within the past 6 months, or New York Heart Association [NYHA] functional class III-IV);
  3. Uncontrolled epilepsy, severe psychiatric disorders, or a history of severe psychiatric disorders;
  4. History of organ transplantation;
  5. Diabetes mellitus or hypertension that is not adequately controlled;
  6. Presence of autoimmune diseases, immune-related extrahepatic manifestations (including vasculitis, purpura, polyarteritis nodosa, peripheral neuropathy, and glomerulonephritis), thyroid diseases, malignancies, or receipt of immunosuppressive therapy;
  7. Presence of serious underlying diseases such as severe infection, heart failure, chronic obstructive pulmonary disease, or other serious diseases;
  8. History of alcohol abuse or drug addiction.
* Total bilirubin > 51 μmol/L, or serum albumin < 28 g/L, or prothrombin time prolonged by > 6 seconds;
* Creatinine clearance<60mL/min；
* Co-infection with hepatitis A, C, or E virus, or HIV infection;
* Use of interferon within 3 months prior to screening;
* Positive pregnancy test in female subjects;
* Abnormal hematology results: white blood cell count (WBC) < 3×10^9/L, neutrophil count 1.5×10^9/L, or platelet count 60×10^9/L；
* Current use of prohibited medications that cannot be discontinued;
* Use of L47 or Myrcludex B within 3 months prior to screening;
* Subjects receiving standardized nucleos(t)ide analogue (NA) therapy with a treatment duration of less than 12 weeks;
* Other significant abnormalities in laboratory tests or auxiliary examinations that, in the opinion of the investigator, make the subject unsuitable for participation in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who achieved response | 48 weeks of treatment
  HDV RNA suppression (< LLOQ) or a decrease of ≥ 2 log10 from baseline combined with ALT normalization

SECONDARY OUTCOMES:
Proportion of subjects with a ≥ 2 log₁₀ decrease in HDV RNA from baseline | 48 weeks of treatment
Proportion of subjects with a ≥ 2 log₁₀ decrease in HDV RNA from baseline and normalized ALT | Continuous treatment for 48 weeks
Proportion of subjects with HDV RNA below the limit of detection (LOD) | Continuous treatment for 48 weeks
Changes in HDV RNA relative to baseline | Continuous treatment for 48 weeks
Proportion of subjects with normalized ALT | Continuous treatment for 48 weeks
Changes in ALT relative to baseline | Continuous treatment for 48 weeks
Changes in HBV-related parameters (HBV DNA, HBeAg, qHBsAg, etc.) | Continuous treatment for 48 weeks
Changes in histological response of the liver | Continuous treatment for 48 weeks
Change in Model for End-Stage Liver Disease (MELD) score | Continuous treatment for 48 weeks
Change in Child-Turcotte-Pugh score | Continuous treatment for 48 weeks
Occurrence of liver-related endpoint events | continuous treatment for 48 weeks
  such as cirrhosis, hepatic decompensation, HCC, liver transplantation / liver-related death, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Junqi Niu, Professor, Study Chair — The First Hospital of Jilin University; Yanhang Gao, Study Chair — The First Hospital of Jilin University
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No